CLINICAL TRIAL: NCT05252962
Title: Investigation of the Bioavailability of Marine Based Collagen Peptides in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rousselot BVBA (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BTS1786/21
Record Dates: First submitted 2022-02-01; First posted 2022-02-23 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: The clinical study will be performed in a double-blind, randomized, monocentric cross-over design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- marine collagen peptide production process I (Experimental): standardized to 10 g provided as single dose. Orally applied in water.
  Interventions: Dietary Supplement: Collagen Peptides
- marine collagen peptide production process II (Experimental): standardized to 10 g provided as single dose. Orally applied in water.
  Interventions: Dietary Supplement: Collagen Peptides
- marine collagen peptide fish source I (Experimental): standardized to 10 g provided as single dose. Orally applied in water.
  Interventions: Dietary Supplement: Collagen Peptides
- marine collagen peptide fish source II (Experimental): standardized to 10 g provided as single dose. Orally applied in water.
  Interventions: Dietary Supplement: Collagen Peptides

INTERVENTIONS:
Dietary Supplement: Collagen Peptides — Collagen peptides will be orally administered and pharmacokinetic parameters will be assessed up to 6 hours after study product intake.

SUMMARY:
The aim of this study is to evaluate the relative bioavailability of Peptan® Type I collagen peptides from different marine origin (different fish sources, production process and molecular weight) in healthy human subjects.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the relative bioavailability of different Peptan® Type I collagen peptides in healthy human subjects. The pharmacokinetic parameters AUC0-6h, Cmax and Tmax will be determined from the concentration-time curves of characteristic collagen markers (e.g. hydroxyproline, proline, glycine, di- and tripeptides together with further amino acids) after oral single dose administration.

The following objectives will be evaluated by comparison of pharmacokinetic parameters between the products:

* The impact of different production processes
* The impact of size of collagen peptides
* The impact of different fish sources

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations
* Age: 18 - 50 years
* Healthy men and women
* BMI: 19 - 28 kg/m2
* Non-smoker

Exclusion Criteria:

* Relevant history or presence of any severe medical disorder, potentially interfering with this study (e.g. mal absorption, chronic gastro-intestinal diseases, heavy depression, diabetes, acute cancers within last 3 years except basal cell carcinoma of the skin, etc.)
* A significant CVD event within last 3 mo. incl. myocardial infarction, stroke, congestive heart failure
* Significant changes in lifestyle or medication (within last 3 mo.) or surgical intervention or surgical procedure such as bariatric surgery
* For this study clinically relevant abnormal laboratory, ECG, vital signs or physical findings at screening
* Blood donation within 1 month prior to study start or during study
* "Extreme dietary regimes": vegan lifestyle, weight loss diet with <1200 kcal/day for women and <1800 kcal for men
* Intake of anticoagulants like Heparin, Marcumar etc.
* Regular intake of drugs or supplements possibly interfering with this study within 2 weeks prior to study start or during study
* History of hypersensitivity to fish

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC(0-6h)) for hydroxyproline after single dose of the different collagen peptides. | pre dose and up to 6 hours post dose
  Pharmakokinetic variable
Peak plasma concentration after administration (Cmax) for hydroxyproline after single dose of the different collagen peptides. | pre dose and up to 6 hours post dose
  Pharmakokinetic variable
Time to reach the maximum concentration of hydroxyproline (Tmax) for hydroxyproline after single dose of the different collagen peptides. | pre dose and up to 6 hours post dose
  Pharmakokinetic variable

SECONDARY OUTCOMES:
Area Under the Curve (AUC(0-6h)) of other characteristic amino acids, total amino acids, as well as the selected di- and tripeptides | pre dose and up to 6 hours post dose
  Pharmakokinetic variables
Peak plasma concentration after administration (Cmax) of other characteristic amino acids, total amino acids, as well as the selected di- and tripeptides | pre dose and up to 6 hours post dose
  Pharmakokinetic variables
Time to reach the maximum concentration (Tmax) of other characteristic amino acids, total amino acids, as well as the selected di- and tripeptides | pre dose and up to 6 hours post dose
  Pharmakokinetic variables

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Virgilio, PhD, Study Director — RousselotBVBA
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany